CLINICAL TRIAL: NCT02520557
Title: An Exploratory Case-Control Study of Genetic and Clinical Factors for Serious Cutaneous Reactions Among Users of Eslicarbazepine Acetate
Brief Title: An Exploratory Study of Genetic and Clinical Factors for Serious Skin Reactions Among Users of Eslicarbazepine Acetate
Status: Terminated | Type: Observational
Why Stopped: The study was not terminated for safety reasons. The sponsor was released from the postmarketing requirement to conduct the study
Sponsor: Sumitomo Pharma America, Inc. (Industry)
Collaborators: University of Pennsylvania (Other)
Responsible Party: Sponsor
Other Study IDs: SEP093-452
Record Dates: First submitted 2015-08-04; First posted 2015-08-13 (Estimated); Last update posted 2021-01-22 (Actual); Status verified 2021-01

CONDITIONS: SCAR
Keywords: Epilepsy; Genetic associations with severe Cutaneous Adverse Reactions
MeSH Terms: conditions — Cicatrix; Epilepsy | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Blood or Saliva
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Case: Cases will be individuals with documented definite or probable Stevens-Johnson syndrome (SJS), toxic epidermal necrolysis (TEN), acute generalized exanthematous pustulosis (AGEP), or drug reaction with eosinophilia and systemic symptoms (DRESS) or symptom onset consistent with one of these conditions within the first 4 months of using ESL (including up to 14 days after discontinuing ESL) will be considered a potential case. Blood draw or Saliva.
  Interventions: Other: Blood or Saliva
- Control: Controls will be individuals who have used ESL for at least 6 weeks and who have not developed SCAR. Blood draw or saliva.
  Interventions: Other: Blood or Saliva

INTERVENTIONS:
Other: Blood or Saliva — To screen for HLA genotypes that may place patients at high risk of SCAR when they use ESL.

SUMMARY:
The reason for this study is to understand if people with certain genes are predisposed to develop severe skin reactions after they are administered Eslicarbazepine Acetate. Currently there is no information that suggests that certain individuals who use Eslicarbazepine Acetate are predisposed to develop severe skin reactions. However, previous research has shown that seizure medicines like carbamazepine (Tegretol®) and oxcarbazepine (Trileptal®, Oxtellar XR®) are more likely to cause severe drug related skin reactions in some people of Asian ancestry who have specific genes. These are genes found in an area of chromosomes called the Major Histocompatibility Complex. This association is called a genetic risk factor. The study objective is to compare information that is obtained from individuals with a history of seizure disorders who develop severe skin reactions while using Eslicarbazepine Acetate to a group of patients who also have a history of seizure disorders and do not have a history of a severe skin reaction after using Eslicarbazepine Acetate.

DETAILED DESCRIPTION:
This study is a genetic case-control study conducted in the United States. In case-control studies, cases with a condition of interest (in this case, individuals with SCAR [severe cutaneous adverse reactions] after initiating ESL); and controls, individuals known to not have the condition of interest (in this case ESL users without SCAR), are identified. Cases will be individuals with documented definite or probable Stevens-Johnson syndrome (SJS), toxic epidermal necrolysis (TEN), acute generalized exanthematous pustulosis (AGEP), drug reaction with eosinophilia and systemic symptoms (DRESS) or symptom onset consistent with one of these conditions within the first 4 months of using ESL (including up to 14 days after discontinuing ESL), ascertained through PPD Pharmacovigilance (PVG) (Sponsor CRO). Controls will be individuals who have used ESL for at least 6 weeks but did not develop any SCAR and will be matched by genetic ancestry classification in a ratio of up to 10 controls per case. Controls will be collected prospectively, so that a pool of ESL-tolerant patients will be identified independently of the collection of cases. Controls will be selected from among:

* Ongoing subjects in clinical studies of ESL; and
* Patients prescribed ESL who may be asked to participate by neurologists at high-prescribing practices with high ethnic diversity.

Blood or saliva samples for genotyping ancestry markers (for matching controls to cases) and sequencing the HLA regions will be collected from cases and control subjects after they have provided consent for participation in a genetic study. In addition, a blood sample will be requested from subjects to assess the relationship with specific viral markers.

ELIGIBILITY:
Inclusion Criteria:

* Study subjects must have the ability to comprehend the informed consent and be willing to provide informed consent and consent for storage and DNA testing of blood or saliva. For subjects who are unable to comprehend the written consent, a legal guardian who is able to describe and provide an understanding of the informed consent to the subject must sign all study consent forms on behalf of the subject.
* The study subject or parent/guardian must possess an educational level and degree of understanding of English or Spanish that enables them to communicate suitably with the local investigator and study coordination staff.

Specific criteria for cases and controls:

* Cases will be individuals with documented definite or probable Stevens-Johnson syndrome (SJS)
* Toxic epidermal necrolysis (TEN), acute generalized exanthematous pustulosis (AGEP), or drug reaction with eosinophilia and systemic symptoms (DRESS)
* Symptom onset consistent with one of these conditions within the first 4 months of using ESL (including up to 14 days after discontinuing ESL).
* Controls will be individuals who have used ESL for at least 6 weeks and who have not developed SCAR.

Exclusion Criteria:

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Males and Females with a history of seizure disorders who may or may not develop severe skin reactions while using Eslicarbazepine
Sampling Method: Probability Sample
Enrollment: 121 (Actual)
Dates: Start 2015-11-30 (Actual); Primary Completion 2020-01-21 (Actual); Study Completion 2020-01-21 (Actual)

PRIMARY OUTCOMES:
Severe Cutaneous Adverse Reactions (SCAR) while using ESL | up to 4 months

SECONDARY OUTCOMES:
HLA genotypes that may place patients at high risk of SCAR when they use ESL. | up to 4 months

CONTACTS AND LOCATIONS:
Overall Officials: CNS Medical Director, Study Director — Sumitomo Pharma America, Inc.
Locations (1):
- University of Pennsylvania Perlman School of Medicine, Philadelphia, Pennsylvania, United States